CLINICAL TRIAL: NCT04940975
Title: Effectiveness of an Occupation-based Sleep Program for People With Insomnia
Brief Title: Occupation-based Sleep Program for People With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20180610001
Record Dates: First submitted 2021-03-05; First posted 2021-06-28 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-03

CONDITIONS: Insomnia, Primary; Insomnia
Keywords: Insomnia; Occupational Therapy; Sleep; Evaluation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupation-based sleep intervention program (Experimental): A program composed of four occupation-based interactive workshops on sleep, insomnia, lifestyle, and change strategies, plus two individual coaching sessions on lifestyle and sleep hygiene.
  Interventions: Behavioral: Occupation-based sleep intervention program
- Insomnia educational program (Treatment as Usual Group) (Active Comparator): A program composed of four educational talks on sleep hygiene and relaxation training, plus two individual sessions for the reviewing of sleep patterns.
  Interventions: Behavioral: Insomnia Education Program at Integrated Mental Health Clinic (IMHC)

INTERVENTIONS:
Behavioral: Occupation-based sleep intervention program — A program composed of four occupation-based interactive workshops on sleep, insomnia, lifestyle, and change strategies, plus two individual coaching sessions on lifestyle and sleep hygiene.
  Arms: Occupation-based sleep intervention program
Behavioral: Insomnia Education Program at Integrated Mental Health Clinic (IMHC) — A program composed of four educational sessions on sleep and insomnia, plus relaxation training, plus two individual review sessions on sleep hygiene with participant.
  Arms: Insomnia educational program (Treatment as Usual Group)

SUMMARY:
Introduction. Sleep problems are a health issue worldwide. Based on the Person-Environment-Occupation-Performance model and the theory of occupational balance, we developed an occupation-based sleep program to address several objectives by lifestyle intervention: 1) minimize the influence of bodily function on sleep; 2) promote an environment conductive to sleep; and 3) restructure daytime activity with a focus on occupational balance through psychoeducation and lifestyle coaching.

Method. This study aims to evaluate the effectiveness of an occupation-based sleep intervention on sleep pattern, mood, and occupational balance among community-dwelling adults with insomnia when compared with other, more usual, forms of treatment, typically focused on education, sleep hygiene, and relaxation. A total of 42 subjects were recruited: 22 for the intervention group and 20 for the treatment as usual group.

DETAILED DESCRIPTION:
The goal of this study is to investigate the effectiveness of occupation-based sleep program for patients with insomnia. It compares the treatment outcomes of sleep pattern, mood, and occupational balance between an intervention group (occupation-based sleep program) and a treatment-as-usual (TAU) group (sleep hygiene education and relaxation training) upon completion of their respective programs and at one-month follow up.

The occupation-based sleep program includes both group and individual sessions. Each group consists of 4 to 6 patients. Each session last for two hours and are held on a weekly basis. Group session focus on sharing information and goal setting to facilitate the formation of good habits and positively restructure lifestyle. Individual coaching sessions aim to follow up on action planning to promote occupational balance.

This study uses a quasi-experimental design. The participants of the intervention group attended the occupation-based sleep program in general outpatient clinic A. Participants in the comparison group received TAU in a general outpatient clinic B of another district. The three time-points for collection of outcome data are at baseline (T1), after the intervention (week 8) (T2), and a one-month post intervention follow up (week 12) (T3). The outcomes will be collected by a blinded assessor who is not involved in the delivery or administration of the study.

Participants The inclusion criteria for recruitment of participants are: 1) diagnosis of insomnia disorder, 2) referral by general practitioner; 3) aged 18 to 65 years old; 4) Insomnia Severity Index score over 14; 5) regularly uses a smart phone, which enable data synchronization with the MiBand2 activity wristband; 6) able to complete self-administered study questionnaires and 7) able to communicate in Cantonese. The exclusion criteria are: 1) diagnosis of severe mental illness; 2) Personal Health Questionnaire 9 (measures depressive symptoms), score over 19 and/or anxiety symptoms (General Anxiety Disorder 7 score over 15); 3) On regular pain medication during the last month, for more than 3 days per week); 4) sleep affected by respiratory disease or 5) regular user of alcohol or addictive substances.

Instruments

The primary outcome measures of the study are insomnia and sleep quality, and the secondary measures are measures of occupational balance, depression, and anxiety.

Cantonese Version Insomnia Severity Index (C-ISI). The C-ISI is a self-report questionnaire that measures the severity of insomnia. A higher score indicate more severe insomnia: Total of 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe). Previous studies have reported adequate psychometric properties for both the English and Chinese versions. Reliability is excellent (α = 0.90-0.91). Sensitivity and specificity at cut-off 10 were 86.1% and 87.7%, respectively.

Chinese Version Pittsburgh Sleep Quality Index (C-PSQI). The C-PSQI is a self-report questionnaire that measures sleep quality. The questions focus on seven aspects of sleep: 1) quality; 2) latency; 3) duration; 4) efficiency; 5) disturbance; 6) use of sleep medication; 7) daytime dysfunction. Under the seven component scores, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.The psychometric properties of the PSQI have been well documented. The Chinese translated version demonstrated good internal consistency (α = 0.82-0.83), and acceptable test-retest reliability over a 14- to 21-day intervals (r = 0.77) for patient with insomnia. It demonstrated good convergent validity, with significant correlations with sleep quality-visual analogues scale and sleep diary. It could differentiate people with and without insomnia, sensitive and specificity of 98% and 55% respectively.

Activity Wristband. The Mi Band 2 is a commercially available activity wristband commonly used for measuring activity level and sleep pattern. A recent research stated that three types of CAM (including Mi Band 2, the device selected for use in the present study) were good at detecting the most basic parameters, actual time spent in bed. MiBand2 that was selected for this study monitors a user's sleep and physical activity neutrally. It provides objective data on sleep duration on a weekly basis, including information about sleep duration, number of nighttime awakenings, and typical sleeping habits.

Occupational Balance Questionnaire (OB-Quest). The OB-Quest is a self-completed questionnaire developed to measure occupational balance in daily life, It focuses on satisfaction with the amount and variation of occupation. It consists of 13 items measured on six-step ordinal scales, and a lower score indicates a better balance. The internal consistency of the OB-Quest is 0.9, and test-retest reliability is also 0.9. A translation and validation study of the Chinese OB-Quest was completed. The study results showed that the Chinese version of OB-Quest can be readily used for research with Chinese persons.

Personal Health Questionnaire 9 (PHQ9). PHQ9 is a self-administered version of part of the Primary Care Evaluation of Mental Disorders (PRIME-MD) diagnostic instrument for common mental disorders. It is the depression module of the PHQ, which scores each of the nine Diagnostic & Statistical Manual version 4 (DSM-IV) criteria as "0" (not at all) to "3" (nearly every day). It has been validated for use in primary care, for monitoring the severity of depression and response to treatment. A higher total score indicate more severe depression. It is commonly used for screening depression. PHQ9 is a reliable tool with good reliability and validity. The psychometric properties for patients with depression in a Chinese primary care population were found to be acceptable to good.

d General Anxiety Disorder-7 (GAD 7). This questionnaire is part of the PRIME-MD diagnostic instrument for common mental disorders. The Generalised Anxiety Disorder-7 (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks.

The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and ' nearly'. The Cut points of 5, 10, and 15 might be interpreted as representing mild, moderate, and severe levels of anxiety on the GAD-7. Previous studies have shown GAD7 to have a high degree of reliability and validity, as well as high internal consistency.

Statistical Analysis The Statistical Package for the Social Sciences (SPSS) (Version 25) is used for data analysis. Descriptive statistics were used to describe the demographic characteristics and outcomes. The baselines of the two groups were compared by t test and Chi-square. Repeated measure ANOVA (General Linear Model) was used to analyze the effectiveness of the program. Pairwise difference was tested on the outcomes between different time points (baseline vs. post treatment, post treatment vs. one-month follow-up), between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of insomnia disorder
* Referral by general practitioner
* Aged 18 to 65 years old
* Insomnia Severity Index score over 14
* Regularly uses a smart phone, which enable data synchronization with the MiBand2 activity wristband
* Able to complete self-administered study questionnaires
* Able to communicate in Cantonese

Exclusion Criteria:

* Diagnosis of severe mental illness
* Personal Health Questionnaire 9 (measures depressive symptoms), score over 19 and/or anxiety symptoms (General Anxiety Disorder 7 score over 15);
* On regular pain medication during the last month, for more than 3 days per week
* Sleep affected by respiratory disease
* Regular user of alcohol or addictive substances.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Cantonese Version Insomnia Severity Index (C-ISI) | Baseline
  self-report questionnaire that measures the severity of insomnia. The score range from 0-28. A higher score indicate more severe insomnia
Cantonese Version Insomnia Severity Index (C-ISI) | Post (8th week)
  self-report questionnaire that measures the severity of insomnia. The score range from 0-28. A higher score indicate more severe insomnia
Cantonese Version Insomnia Severity Index (C-ISI) | Follow-up (12th week)
  self-report questionnaire that measures the severity of insomnia. The score range from 0-28. A higher score indicate more severe insomnia
Chinese Version Pittsburgh Sleep Quality Index (C-PSQI). | Baseline
  self-report questionnaire that measures sleep quality. The total scores range from 0 to 21. Higher scores indicate worse sleep quality.
Chinese Version Pittsburgh Sleep Quality Index (C-PSQI). | Post (8th week)
  self-report questionnaire that measures sleep quality. The total scores range from 0 to 21. Higher scores indicate worse sleep quality.
Chinese Version Pittsburgh Sleep Quality Index (C-PSQI). The total scores range from 0 to 21. Higher scores indicate worse sleep quality. | Follow-up (12th week)
  self-report questionnaire that measures sleep quality.
MiBand2 Activity Wristband. | Baseline
  commercial activity monitor (CAM) commonly used for measuring activity level and sleep pattern. There is no definite range for activity level and sleep pattern, but higher activity level and shorter sleep duration indicates a poorer sleep pattern.
MiBand2 Activity Wristband. | Post (8th Week)
  commercial activity monitor (CAM) commonly used for measuring activity level and sleep pattern. There is no definite range for activity level and sleep pattern, but higher activity level and shorter sleep duration indicates a poorer sleep pattern.
MiBand2 Activity Wristband. | Follow-up (12th week)
  commercial activity monitor (CAM) commonly used for measuring activity level and sleep pattern. There is no definite range for activity level and sleep pattern, but higher activity level and shorter sleep duration indicates a poorer sleep pattern.

SECONDARY OUTCOMES:
Occupational Balance Questionnaire (OB-Quest) | Baseline
  measure occupational balance and lifestyle in daily life. The total score ranges from 10-30, and a higher score indicates a poorer balance in occupations.
Occupational Balance Questionnaire (OB-Quest) | Post (8th week)
  measure occupational balance and lifestyle in daily life. The total score ranges from 10-30, and a higher score indicates a poorer balance in occupations.
Occupational Balance Questionnaire (OB-Quest) | Follow-up (12th week)
  measure occupational balance and lifestyle in daily life. The total score ranges from 10-30, and a higher score indicates a poorer balance in occupations.
Personal Health Questionnaire 9 (PHQ9) | Baseline
  commonly used for screening depression. The total score ranges from 0 to 27, and a higher total score indicate more severe depression.
Personal Health Questionnaire 9 (PHQ9) | Post (8th week)
  commonly used for screening depression. The total score ranges from 0 to 27, and a higher total score indicate more severe depression.
Personal Health Questionnaire 9 (PHQ9) | Follow-up (12th week)
  commonly used for screening depression. The total score ranges from 0 to 27, and a higher total score indicate more severe depression.
General Anxiety Disorder 7 (GAD 7). | Baseline
  for screening a range of anxiety disorders in primary care. The total score ranges from 0-21, and a higher score indicates higher anxiety.
General Anxiety Disorder 7 (GAD 7). | Post (8th week)
  for screening a range of anxiety disorders in primary care. The total score ranges from 0-21, and a higher score indicates higher anxiety.
General Anxiety Disorder 7 (GAD 7). | Follow-up (12th week)
  for screening a range of anxiety disorders in primary care. The total score ranges from 0-21, and a higher score indicates higher anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew MH Siu, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - Central Kowloon General Out-Patient Clinic (GOPC), Hong Kong
  - Yau Ma Tai General Out-Patient Clinic (GOPC), Hong Kong

IPD SHARING:
Plan to Share IPD: No